CLINICAL TRIAL: NCT02617433
Title: Relationship Between Muscle Mass Measured by Bioelectrical Impedance Analysis and Muscle Relaxation
Brief Title: Relationship Between Muscle Mass and Muscle Relaxation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Go Eun Bae (Other)
Responsible Party: Sponsor-Investigator, Go Eun Bae, Clinical instructor, Korea University Anam Hospital
Organization: Korea University Anam Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Inbody
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inbody (Experimental): Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Seoul, Korea) after fast for eight hours.
  Interventions: Device: Inbody

INTERVENTIONS:
Device: Inbody — Participant measure muscle mass by bioelectrical impedance analysis (Inbody 720, Seoul, Korea) after fast for eight hours. After measurement, patient is induced anesthesia. Rocuronium dose is 12mg for male, and 9mg for female.

SUMMARY:
Rocuronium block neuromuscular transmission at the neuromuscular junction, causing paralysis of the affected skeletal muscles. There have been several studies reported positive relationship between muscle mass and amount of neuromuscular junction. The purpose of this study is to find relationship between muscle mass and muscle relaxation time.

DETAILED DESCRIPTION:
Rocuronium block neuromuscular transmission at the neuromuscular junction, causing paralysis of the affected skeletal muscles. There have been several studies reported positive relationship between muscle mass and amount of neuromuscular junction. Until now, dose of rocuronium has been judged by patient's weight and height. However, height and weight do not represent exact muscle mass. The purpose of this study is to find relationship between muscle mass and muscle relaxation time. Measurement of muscle mass will be obtained using bioelectrical impedence analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patient who undergo general anesthesia.
* Male; weight 70-75kg , height 170-175cm
* Female; weight 53-58kg , height 158-163cm

Exclusion Criteria:

* Liver and kidney disease
* Any types of muscle disorder.
* Metal materials or pacemaker in body

Ages: 19 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
ratio of result of first stimulus(T1) to result of supramaximal stimulation(T0) | two hours
  T1 and T0 is obtained by train of four which is commonly used neuromuscular monitoring device.

SECONDARY OUTCOMES:
completely suppression time of result of first stimulus(T1). | ten minutes
  T1 is obtained by train of four which is commonly used neuromuscular monitoring device.

OTHER OUTCOMES:
Time until reoccurrence of response of first stimulus(T1). | two hours
  T1 is obtained by train of four which is commonly used neuromuscular monitoring device.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Zhoo Yoon, MD, PhD, Study Director — Korea University Anam Hospital
Locations (1):
- Korea university anam hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided